CLINICAL TRIAL: NCT02731924
Title: Point of Care Ultrasound for Evaluation of Suspected Appendicitis in the Emergency
Brief Title: Point of Care Ultrasound for Evaluation of Suspected Appendicitis in the Emergency Department
Status: Completed | Type: Observational
Sponsor: WellSpan Health (Other)
Collaborators: Stony Brook University (Other)
Responsible Party: Principal Investigator, Brent Becker, Emergency Physician - Wellspan Health York Hospital, WellSpan Health
Other Study IDs: 549570-8
Record Dates: First submitted 2016-04-01; First posted 2016-04-08 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Acute Appendicitis
Keywords: Appendicitis; Ultrasound; Emergency Department
MeSH Terms: conditions — Appendicitis; Emergencies | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ultrasound for Appendicitis: Emergency department patients undergoing point-of-care ultrasound to evaluate for suspected appendicitis
  Interventions: Procedure: Ultrasound for Appendicitis

INTERVENTIONS:
Procedure: Ultrasound for Appendicitis — Point-of-care ultrasound to evaluate emergency department patients for suspected appendicitis

SUMMARY:
The primary purpose of this study is to determine the accuracy of ultrasound (US) in diagnosing appendicitis in emergency department (ED) patients, as compared to the criterion standards of computed tomography, operative reports, or discharge diagnosis.

The secondary purposes of the study include evaluation of the effect of ultrasound for appendicitis on the patient length of stay in the emergency department, the diagnostic utility of specific ultrasound findings in the diagnosis of appendicitis, the role of body mass index (BMI) in the utility of ultrasound for appendicitis and relation of ultrasound findings to the Alvarado score. The study will also examine the inter-rater agreement between point-of- care sonographers' interpretation and blinded reviewers' interpretation of the ultrasound images.

DETAILED DESCRIPTION:
BACKGROUND:

Increasing concerns have been raised over the past several years regarding the degree of radiation exposure in patients being evaluated for abdominal complaints. A deepening body of literature supports the use of ultrasound for the evaluation of appendicitis. In particular, ultrasound is being promoted as first line testing in the evaluation of appendicitis in pediatric populations and adults with BMI < 25. This approach reduces the risks related to radiation exposure and IV contrast dye. Unfortunately, in many practice settings, the availability of radiology-based sonographers is limited and there can be significant delays in obtaining ultrasound images. For these reasons, many ED physicians (EP) have begun to perform bedside ultrasound to evaluate for appendicitis.

Studies have demonstrated a wide range in the accuracy of ultrasound for appendicitis. Sensitivities and specificities vary and no standardized diagnostic criterion exist. Additionally, little has been published directly studying EP point of care ultrasound in the evaluation for acute appendicitis. One study has shown that EP-performed ultrasounds had a relatively low sensitivity, but a high specificity. However, this study was performed by a wide range of users with varying skill levels and older ultrasound machines. The surgical literature suggests that the ability of the clinician to integrate the history, the physical exam and the ultrasound findings in real time improves the diagnostic accuracy of ultrasound for appendicitis.

Currently there are 4 physicians on staff in the ED who are fellowship trained in point of care emergency ultrasound, fully credentialed and are already performing ED based evaluations for appendicitis on a limited basis. The current standard of care is a point of care ultrasound as first-line imaging for patients with suspected appendicitis when a credentialed EP is available to perform the scan. We intend to evaluate the performance of EP-performed point of care ultrasound in the diagnosis of acute appendicitis in ED patients. This study would primarily investigate the accuracy of ultrasound as compared to the criterion standard of either abdominal CT results or surgical pathology report.

STUDY DESIGN:

This will be a prospective, descriptive study of Emergency Department patients suspected of having acute appendicitis. Initial screening of potential enrollees will be performed by ED nurses, residents, and attendings. Once consented and enrolled, a study sonographer will interview and examine the patient, preferably before lab results are available. The ultrasound must be completed and adequate images obtained before other imaging modalities are completed. Ultrasound of the right lower quadrant (RLQ) will performed using the graded compression technique described previously in the literature. All participating EP sonographers are already trained in this technique, fully credentialed and no additional training will be performed. A "Bedside" standardized data collection form will be used at the bedside to record ultrasound findings and clinical information. The sonographer will designate the appendix as "not visualized", "visualized and normal", or "visualized and abnormal" and the ultrasound as "positive for appendicitis", "negative for appendicitis" or "indeterminate" based on the exam and ultrasound findings.

A second sonographer, blinded to all clinical information and the primary sonographer's ultrasound interpretation, will review the de-identified ultrasound images remotely. This overreading sonographer will record his interpretation and secondary findings on a "Blinded Reviewer" standardized data collection sheet.

CT imaging, surgical pathology reports, and a two week telephone follow up will be utilized to determine final outcome of patient's clinical course. At this time, a third "Follow Up" standardized data collection sheet will be used to record patient outcomes and demographic information.

Based on expected proportion of patients with proven appendicitis of 15% with desired precision of 0.15, the estimated sample size for this study is 261.

STUDY POPULATION AND RECRUITMENT METHODS:

Study population will include patients of any age presenting to the emergency department with abdominal pain and a clinical suspicion of appendicitis. Patients will initially be seen by a treating attending physician or resident. If there is a concern for appendicitis the treating physician will contact one of the ultrasound credentialed EP sonographers to perform a point of care ultrasound. Of note, this is the current standard practice in the ED. By choosing to participate in the study, the patient's treatment is not altered in any way from the current standard practice, but simply is agreeing to allow us to collect data and contact them by phone at the two week follow up. The study sonographer will obtain consent. Parental consent will be obtained for patients under the age of 18.

DATA TO BE UTILIZED:

The following data will be recorded:

* Patients initials
* Patient Medical Record Number (MRN)/Financial Identification Number (FIN)
* Age
* Sex
* Height
* Weight
* Symptom Duration
* Chief complaint
* Presence of RLQ pain
* Anorexia
* Migration of pain to RLQ
* Rebound tenderness
* Nausea/vomiting
* Maximum recorded temperature in the Emergency Department
* White Blood Cell (WBC) count
* Visualization of the iliac vessels?
* Visualization of the appendix?
* Maximum outer diameter of the appendix
* Thickness of the appendix wall
* Edema of the wall of the appendix?
* Peri-appendiceal edema or free fluid?
* Non compressible appendix?
* Pain with compression over the appendix?
* Evidence of dilated bowel loops in the RLQ?
* Increased vascularity of the appendix wall?
* Appendicolith?
* Free fluid in the right upper quadrant (RUQ)?
* Diagnostic impression of the sonographer
* Diagnostic impression of the blinded reviewer
* CT diagnosis
* Pathology diagnosis
* Operative report classification
* Time to disposition
* Final diagnosis
* Symptoms/Subsequent diagnosis at two weeks

DATA ANALYSIS:

For the primary outcome, data will be used to calculate the sensitivity and specificity of point of care (POC) US for the diagnosis of appendicitis compared to the criterion standard of CT, operative report, discharge diagnosis and two week follow up phone call.

For secondary outcomes, likelihood ratios for specific ultrasound findings will be determined. Inter-rater agreement between the bedside sonographer and the blinded reviewer will be calculated using Cohen's kappa coefficient. Continuous, time-to-disposition data will be compared utilizing a two-tailed t-test.

Statistical analysis will be performed using SPSS software (IBM, Armonk, NY).

RISKS AND RISK MANAGEMENT:

There are minimal risks to patients participating in this study since ultrasound is non-invasive and known to be safe. There is a slight risk of the participants' privacy or confidentiality being breached. Standard precautions will be taken to ensure privacy and confidentiality is maintained during the study.

BENEFITS:

Patients who have ultrasounds highly suspicious for appendicitis may be referred directly to surgery without further imaging being performed. In these instances study patients would benefit from reduced radiation exposure and faster referral for appropriate surgical care. The results of this study may be used to improve future patient care.

COMPENSATION / INCENTIVES AND RESEARCH-RELATED COSTS:

No compensation will be given to the participants. There will be no research-related costs.

ALTERNATIVE PROCEDURES:

Patients who refuse to participate in the study will not have the quality of their treatment affected in any way.

RESEARCH MATERIALS, METHODS AND CONFIDENTIALITY:

Research records will be stored in locked offices, filing cabinets, and computers using passwords.

SUBJECT INFORMED CONSENT:

We will seek documented informed consent and HIPAA Authorization. ED patients meeting all of the inclusion and exclusion criteria will be asked if they would like to participate in the study by a research sonographer at the time of the ultrasound.

If the patient agrees to participate, the informed consent document will be given to them for their review. If patient declines to participate they will continue their treatment course in the Emergency Department.

REFERENCES:

Burford JM, Dassinger MS, Smith SD. Surgeon-performed ultrasound as a diagnostic tool in appendicitis. Journal of Pediatric Surgery. 2011;46;1115-1120

Estey A, Poonai N, Lim R. Appendix Not Seen: The Predictive Value of Secondary Inflammatory Sonographic Signs. Pediatric Emergency Care. 2013;29(4):435-9.

Fox JC, Solley M, et al. Prospective evaluation of emergency physician performed ultrasound to detect acute appendicitis. European Journal of Emergency Medicine. 2008;15:80-85.

Hulley et al. Designing Clinical Reasearch. 4th ed. Philadelphia, PA: Lippincott, Williams & Wilkins; 2013: Chapter 6.

Karakas SP, Guelfguat M, Leonidas JC, et al. Acute appendicitis in children: comparison of clinical diagnosis with ultrasound and CT imaging. Pediatric Radiology. 2000;30:94-8.

Pacharn P, Ying J, Linam LE, Brody AS, Babcock DS. Sonography in the Evaluation of Acute Appendicitis: Are Negative Sonographic Findings Good Enough? Journal of Ultrasound Medicine. 2010;29;1749-1755.

Puylaert JB. Acute appendicitis: US evaluation using graded compression. Radiology. 1986;158:355-60.

ELIGIBILITY:
Inclusion Criteria:

* RLQ pain with clinical suspicion for acute appendicitis

Exclusion Criteria:

* History of appendectomy
* Imaging prior to ED ultrasound performed to evaluate the RLQ
* Patients who are decisionally impaired or cannot provide consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric emergency department patients at a university-affiliated, community teaching hospital with suspected appendicitis
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Point-of-care Ultrasound for Suspected Appendicitis | 3 years
  The performance of point-of-care ultrasound for appendicitis will be evaluated by comparing each ultrasound to the criterion standard of computed tomography (CT) for each enrolled patient. If a CT is not obtained, then operative report/findings, discharge diagnosis or phone follow up at 2 weeks will be used as the criterion standard to which the ultrasound will be compared.
  Using the criterion standard as the definitive diagnosis for each patient (i.e. presence or absence of appendicitis), each ultrasound will be classified as a true positive, true negative, false positive or false negative. This data will be used to calculated the sensitivity, specificity, likelihood ratios, positive predictive value (PPV), negative predictive value (NPV) and accuracy of point-of-care ultrasound for the diagnosis of appendicitis.

SECONDARY OUTCOMES:
Intraabdominal Free Fluid | 3 years
  The presence or absence of intraabdominal free fluid on ultrasound for appendicitis will be assessed to determine the incidence of this particular sonographic finding in appendicitis, as well as its role in the sonographic diagnosis of appendicitis.
  The sensitivity, specificity and likelihood ratios of this particular sonographic finding in appendicitis will be calculated.
Dilated Loops of Bowel in RLQ | 3 years
  The presence or absence of dilated loops of bowel in the RLQ on ultrasound for appendicitis will be assessed to determine the incidence of this particular sonographic finding in appendicitis, as well as its role in the sonographic diagnosis of appendicitis.
  The sensitivity, specificity and likelihood ratios of this particular sonographic finding in appendicitis will be calculated.
Appendicolith | 3 years
  The presence or absence of an appendicolith on ultrasound for appendicitis will be assessed to determine the incidence of this particular sonographic finding in appendicitis, as well as its role in the sonographic diagnosis of appendicitis.
  The sensitivity, specificity and likelihood ratios of this particular sonographic finding in appendicitis will be calculated.
Appendiceal Dilation | 3 years
  The presence or absence of appendiceal dilation on ultrasound for appendicitis will be assessed to determine the incidence of this particular sonographic finding in appendicitis, as well as its role in the sonographic diagnosis of appendicitis.
  The sensitivity, specificity and likelihood ratios of this particular sonographic finding in appendicitis will be calculated.
Appendiceal Wall Thickening | 3 years
  The presence or absence of appendiceal wall thickening on ultrasound for appendicitis will be assessed to determine the incidence of this particular sonographic finding in appendicitis, as well as its role in the sonographic diagnosis of appendicitis.
  The sensitivity, specificity and likelihood ratios of this particular sonographic finding in appendicitis will be calculated.
Appendiceal Hyperemia | 3 years
  The presence or absence of appendiceal hyperemia on ultrasound for appendicitis will be assessed to determine the incidence of this particular sonographic finding in appendicitis, as well as its role in the sonographic diagnosis of appendicitis.
  The sensitivity, specificity and likelihood ratios of this particular sonographic finding in appendicitis will be calculated.
Inter-rater Agreement | 3 years
  The study will quantify the rate of inter-rater agreement between the clinician performing the point-of-care ultrasound and a blinded reviewer of the ultrasound images.
Patient Length of Stay/Time to Disposition | 3 years
  The study will measure the time to disposition of ED patients undergoing a point of care ultrasound for small bowel obstruction and determine how the ultrasound effects time to patient disposition.
Comparison to Alvarado Score | 3 years
  The study will compare ultrasound findings for appendicitis to diagnostic utility of the Alvarado score in predicting appendicitis.
Body Mass Index | 3 years
  The study will measure the BMI of ED patients and determine how BMI might effect the diagnostic accuracy of point of care ultrasound for appendicitis. BMI cutoff values will be used to define study subgroups for which the sensitivity, specificity and likelihood ratios for appendicitis ultrasound in each subgroup will be calculated and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Brent A Becker, MD, Principal Investigator — Wellspan Health York Hospital
Locations (1):
- Wellspan Health York Hospital, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burford JM, Dassinger MS, Smith SD. Surgeon-performed ultrasound as a diagnostic tool in appendicitis. J Pediatr Surg. 2011 Jun;46(6):1115-20. doi: 10.1016/j.jpedsurg.2011.03.040. PMID 21683208
- [Background] Estey A, Poonai N, Lim R. Appendix not seen: the predictive value of secondary inflammatory sonographic signs. Pediatr Emerg Care. 2013 Apr;29(4):435-9. doi: 10.1097/PEC.0b013e318289e8d5. PMID 23528502
- [Background] Fox JC, Solley M, Anderson CL, Zlidenny A, Lahham S, Maasumi K. Prospective evaluation of emergency physician performed bedside ultrasound to detect acute appendicitis. Eur J Emerg Med. 2008 Apr;15(2):80-5. doi: 10.1097/MEJ.0b013e328270361a. PMID 18446069
- [Background] Hulley et al. Designing Clinical Reasearch. 4th ed. Philadelphia, PA: Lippincott, Williams & Wilkins; 2013: Chapter 6.
- [Background] Karakas SP, Guelfguat M, Leonidas JC, Springer S, Singh SP. Acute appendicitis in children: comparison of clinical diagnosis with ultrasound and CT imaging. Pediatr Radiol. 2000 Feb;30(2):94-8. doi: 10.1007/s002470050023. PMID 10663520
- [Background] Pacharn P, Ying J, Linam LE, Brody AS, Babcock DS. Sonography in the evaluation of acute appendicitis: are negative sonographic findings good enough? J Ultrasound Med. 2010 Dec;29(12):1749-55. doi: 10.7863/jum.2010.29.12.1749. PMID 21098847
- [Background] Puylaert JB. Acute appendicitis: US evaluation using graded compression. Radiology. 1986 Feb;158(2):355-60. doi: 10.1148/radiology.158.2.2934762.
- [Derived] Becker BA, Kaminstein D, Secko M, Collin M, Kehrl T, Reardon L, Stahlman BA. A prospective, multicenter evaluation of point-of-care ultrasound for appendicitis in the emergency department. Acad Emerg Med. 2022 Feb;29(2):164-173. doi: 10.1111/acem.14378. Epub 2021 Sep 14. PMID 34420255